CLINICAL TRIAL: NCT00216476
Title: CONSTATRE: Risperdal Consta Trial Of Relapse Prevention And Effectiveness
Brief Title: A Study of Relapse Prevention and the Effectiveness of Long-acting Injectable Risperidone and Quetiapine Tablets in the Treatment of Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002269
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia, relapse prevention; Antipsychotic agents; Long-acting risperidone; Quetiapine; Aripiprazole
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): Risperidone Long Acting Injectable (LAI) 25 mg injection every 2 weeks until week 104. Dosage may be increased or decreased in steps of 12.5 mg. Additional oral risperidone can be administered as required until a dose increase becomes effective.
  Interventions: Drug: Risperidone Long Acting Injectable (LAI)
- 002 (Active Comparator): Quetiapine Oral tablets are titrated from 50 mg daily to 300-400 mg daily in first 4 days. Subsequently treatment is maintained for 104 weeks and dosage can be adjusted with increments or decrements of 25 to 50 mg.
  Interventions: Drug: Quetiapine
- 003 (Other): Aripiprazole 10-30 mg oral once daily for 104 weeks
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — 10-30 mg oral once daily for 104 weeks
  Arms: 003
Drug: Risperidone Long Acting Injectable (LAI) — 25 mg injection every 2 weeks until week 104. Dosage may be increased or decreased in steps of 12.5 mg. Additional oral risperidone can be administered as required until a dose increase becomes effective.
  Arms: 001
Drug: Quetiapine — Oral tablets are titrated from 50 mg daily to 300-400 mg daily in first 4 days. Subsequently treatment is maintained for 104 weeks and dosage can be adjusted with increments or decrements of 25 to 50 mg.
  Arms: 002

SUMMARY:
The purpose of this study is to investigate whether a long-acting injectable formulation of risperidone provides better effectiveness over 2 years, as measured by the time to relapse, compared with quetiapine tablets in a routine psychiatric care setting. Aripiprazole will be investigated in a descriptive manner.

DETAILED DESCRIPTION:
Although many schizophrenia patients currently take oral antipsychotic medications, it is estimated that up to 75% of them have difficulty adhering to the daily oral regimen. Long-acting injectable formulations may eliminate the need for daily medication and enhance patient compliance with the treatment regimen. This is an open-label (all people involved know the identity of the intervention), randomized (study drug assigned by chance) study of a formulation of risperidone (coated microspheres) injected into the muscle at 2 week intervals over 104 weeks in stable patients with schizophrenia or schizoaffective disorder, who are being treated with oral risperidone, olanzapine, or other conventional antipsychotic agents. A comparator group will receive tablets of quetiapine to be taken 2 or 3 times daily, depending on the optimal dosage. In countries where aripiprazole is available, aripiprazole was also included in a descriptive manner. Reasons for switching symptomatically stable patients from their current antipsychotic treatment include insufficient effectiveness of the medication on symptoms, adverse events, or a patient's request. The principal measure of effectiveness of the drug is the time to relapse. Assessments of effectiveness also include: Positive and Negative Syndrome Scale (PANSS), which measures the symptoms of schizophrenia; overall severity of illness measured by the Clinical Global Impression subscale (CGI-S); patient's condition measured by the Clinical Global Impression condition subscale (CGI-C); quality of life assessed by the SF-12 survey. Safety evaluations include incidence of adverse events, Extrapyramidal Symptoms Rating Scale (ESRS), clinical laboratory tests (biochemistry, haematology, and urinalysis), and vital signs (pulse, blood pressure). The study hypothesis is that treatment with long-acting risperidone injected intramuscularly every 2 weeks provides better effectiveness than quetiapine, as measured by time to relapse, in patients with schizophrenia or schizoaffective disorder. Risperidone injections 25mg biweekly for 104 weeks, increasing or decreasing (increments of 12.5mg) at investigator's discretion. Risperidone tablets (2mg daily for 2 days) for patients starting on risperidone. Quetiapine and Aripiprazole used according to package insert.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV)
* Patients currently treated with oral risperidone, olanzapine or a conventional neuroleptic monotherapy at doses not exceeding 6 mg risperdal, 20 mg olanzapine, or a conversion dose of 10 mg haloperidol for oral conventional agents
* Patients who are stable (judged clinically stable by the investigator and on a stable dose of medication for 4 weeks or longer) but not optimally treated (non-satisfactory treatment regarding symptoms or adverse events)

Exclusion Criteria:

* Diagnosis other than schizophrenia or schizoaffective disorder by DSM-IV Axis I criteria
* Patients being treated with antipsychotic agents other than oral risperidone, olanzapine or conventional oral neuroleptic agents
* Patients with known hypersensitivity to oral risperidone, quetiapine, aripiprazole, or who are known non-responders to oral risperidone, quetiapine, aripiprazole or to previous treatment with at least 2 antipsychotic agents
* Patients treated with mood stabilizers or antidepressants who are not on stable dose for at least 3 months before study initiation
* Pregnant or nursing females, or those lacking adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 753 (Actual)
Dates: Start 2004-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (96):
- Austria (3):
  - Hall in Tirol
  - Linz
  - Neunkirchen
- Bulgaria (3):
  - Pleven
  - Sofia
  - Sofia Sofia
- Croatia (4):
  - Osijek
  - Rijeka
  - Split
  - Zagreb
- Czechia (9):
  - Brno
  - Lnáře
  - Opava
  - Pardubice
  - Plzen Czechia
  - Prague
  - Praha 2 N/A
  - Uherský Brod
  - Ústí nad Labem
- Denmark (2):
  - Middelfart
  - Vordingborg
- Estonia (3):
  - Pÿrnu N/A
  - Tallinn
  - Tartu
- France (10):
  - Bron
  - Brumath
  - Créteil
  - Dieppe
  - Hénin-Beaumont
  - Mont-Saint-Martin
  - Poitiers
  - Reims
  - Roubaix
  - Toulouse
- Germany (10):
  - Augsburg
  - Berlin
  - Bochum
  - Duisburg
  - Düsseldorf
  - Karlstadt am Main
  - Krefeld
  - München
  - Oranienburg
  - Stralsund
- Greece (2):
  - Heraklion -Crete
  - Thessalonikis
- Hungary (6):
  - Budapest
  - Gyõr
  - Gyula
  - Kistarcsa
  - Szeged
  - Vác
- Ireland (4):
  - Cork
  - Dublin
  - Kerry
  - Sligo
- Israel (3):
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- Latvia (2):
  - Jelgava
  - Riga
- Lithuania (5):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Poland (4):
  - Choroszcz
  - Gdynia Na
  - Poznan
  - Warsaw
- Portugal (2):
  - Coimbra
  - Porto
- Romania (3):
  - Bucharest
  - Craiova
  - Iași
- Khobar, Saudi Arabia
- Slovakia (2):
  - Košice
  - Zvolen
- Slovenia (3):
  - Begunje na Gorenjskem
  - Ljubljana
  - Ormož
- Spain (4):
  - Madrid
  - Oviedo (Asturias)
  - Seville
  - Valencia
- Sweden (2):
  - Gothenburg
  - Trollhättan
- Turkey (Türkiye) (4):
  - Ankara Turkey
  - Bakirkoy/Istanbul N/A
  - Istanbul
  - Izmir
- United Kingdom (5):
  - Barnet
  - Barnsley
  - Hull
  - Llantrissant
  - Swansea

REFERENCES:
- See also: CONSTATRE: Risperdal� Consta� Trial of Relapse Prevention and Effectiveness RIS-SCH-3001 Study Results Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=46&filename=CR002269_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects had a diagnosis of schizophrenia or schizoaffective disorder (according to the Diagnostic and Statistical Manual of Mental Disorders - 4th edition [DSM-IV]) and were treated with oral risperidone, olanzapine, or conventional oral neuroleptic monotherapy at screening. They were to be symptomatically stable but not optimally treated.
Groups:
- Risperidone LAI: Risperidone Long Acting Injectable (LAI) intramuscular injection, dose of 25, 37.5, or 50 mg every 2 weeks
- Quetiapine: oral Quetiapine, target dose of 300-400 mg twice daily (b.i.d.) or three times daily (t.i.d.)
- Aripiprazole: oral Aripiprazole, recommended maintenance dose of 10-30 mg once daily (q.d.)
Period: Overall Study
Arm/Group | Risperidone LAI | Quetiapine | Aripiprazole
Started | 329 | 337 | 45
Completed | 224 | 230 | 28
Not Completed | 105 | 107 | 17
Not completed — Withdrawal by Subject | 59 | 72 | 9
Not completed — Lost to Follow-up | 10 | 9 | 1
Not completed — Adverse Event | 6 | 10 | 1
Not completed — Lack of Efficacy | 4 | 3 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1
Not completed — Refuses Injection | 11 | 0 | 0
Not completed — No Further Need for Treatment | 3 | 4 | 1
Not completed — Non-compliance | 0 | 4 | 1
Not completed — Higher dose/Extra Medication Required | 2 | 0 | 2
Not completed — Administrative Reasons | 1 | 1 | 0
Not completed — Protocol Deviation | 5 | 1 | 0
Not completed — Patient Moved | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Risperidone LAI: intramuscular injection, dose of 25, 37.5, or 50 mg every 2 weeks
- Quetiapine: oral, target dose of 300-400 mg b.i.d. or t.i.d.
- Total: Total of all reporting groups
Arm/Group | Risperidone LAI | Quetiapine | Total
Number analyzed (Participants) | 329 | 337 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] — As aripiprazole was not part of the primary analysis but was only added for exploratory purposes, data on this arm are not presented here.
  years | 40.6 (12.48) | 42.6 (13.14) | 41.6 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants] — As aripiprazole was not part of the primary analysis but was only added for exploratory purposes, data on this arm are not presented here.
  Participants
    Female | 134 | 146 | 280
    Male | 195 | 191 | 386
Race/Ethnicity, Customized [Number; unit: participants] — As aripiprazole was not part of the primary analysis but was only added for exploratory purposes, data on this arm are not presented here.
  participants
    Caucasian | 320 | 330 | 650
    Oriental | 1 | 2 | 3
    Hispanic | 2 | 0 | 2
    Black | 1 | 0 | 1
    Arab | 5 | 4 | 9
    Pakistani | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — As aripiprazole was not part of the primary analysis but was only added for exploratory purposes, data on this arm are not presented here.
  kg/m2 | 27.6 (5.23) | 27.0 (5.32) | 27.3 (5.28)
Weight [Mean (Standard Deviation); unit: kg] — As aripiprazole was not part of the primary analysis but was only added for exploratory purposes, data on this arm are not presented here.
  kg | 80.4 (16.93) | 79.0 (17.75) | 79.7 (17.35)

OUTCOME MEASURES:

1. Primary Outcome: Mean Relapse Free Period(Risperidone LAI Versus Quetiapine)
Description: Relapse was defined as meeting any of the predefined criteria (adapted from Csernansky et al., 2002) on 2 consecutive evaluations during treatment, 3 to 5 days apart. The relapse rate in each treatment arm was estimated using the Kaplan-Meier method.
Time Frame: Assessed at each visit from the moment the subject was randomized to a treatment arm (baseline visit) until the end of treatment (Week 104 or earlier)
Population: Efficacy analysis set, defined as all subjects who received at least 1 dose of study medication and who had at least 1 efficacy assessment after baseline. This excluded 2 subjects of the risperidone LAI arm and 11 of the quetiapine arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Risperidone LAI | Quetiapine
Number analyzed (Participants) | 327 | 326
days | 607 (11.4) | 533 (15.6)
Statistical Analysis 1: Comparison: Risperidone LAI vs Quetiapine; Null hypothesis was that there is no difference in treatment effect between risperidone LAI and quetiapine by mean relapse free period; given a estimated relapse rate of 30% for risperidone LAI and 42% for quetiapine, with 80% power and 5% 2-tailed significance level, 251 subjects were needed per treatment arm. To adjust for an estimated 20% discontinuations for reasons other than relapse, 628 subjects in total were needed. Actual relapse rates were 17% (risperidone LAI) and 31% (quetiapine); Test type: Superiority or Other; p < 0.0001, Log Rank — threshold for significance: 0.05 (2-sided)

2. Secondary Outcome: Mean Relapse Free Period (Exploratory/Aripiprazole)
Description: As for risperidone and quetiapine, relapse was defined as meeting any of the predefined criteria (adapted from Csernansky et al., 2002) on 2 consecutive evaluations during treatment, 3 to 5 days apart. Since aripiprazole was new on the market at the time the study was conducted, this aripiprazole analysis was exploratory.
Time Frame: as for outcome 1
Population: Efficacy analysis set, defined as all subjects who received at least 1 dose of study medication and who had at least 1 efficacy assessment after baseline. This excluded 1 subject of the aripiprazole arm.
Measure: Mean (Standard Error); unit: days
Groups:
- Aripiprazole: oral, recommended maintenance dose of 10-30 mg q.d.
Arm/Group | Aripiprazole
Number analyzed (Participants) | 44
days | 314 (20.4)

3. Secondary Outcome: Change From Baseline to Endpoint in Total Positive and Negative Syndrome Scale (PANSS) Score
Description: The neuropsychiatric symptoms of schizophrenia were assessed by means of the 30-item PANSS scale. The PANSS scale provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, i.e., the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items).
  Each item of the scale is to be scored on a scale of 1 (absent) to 7 (extreme).
Time Frame: as for outcome 1
Population: Efficacy analysis set, defined as all subjects who received at least 1 dose of study medication and had at least 1 efficacy assessment after baseline. This excluded 2 subjects of the risperidone LAI, 11 of the quetipaine, and 1 of the aripiprazole arm. One additional subject in each the risperidone LAI and quetiapine arm did not have PANSS data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone LAI | Quetiapine | Aripiprazole
Number analyzed (Participants) | 326 | 325 | 44
units on a scale | -9.3 (25.65) | -1.1 (26.28) | -7.7 (27.99)
Statistical Analysis 1: Comparison: Risperidone LAI vs Quetiapine; Between-group comparison of the change from baseline to endpoint in total PANSS score. The endpoint of the study was based on the Last Observation Carried Forward (LOCF) principle, i.e., it was defined as the last available visit during the study with non-missing data for a parameter (excluding the baseline value); Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — The statistical test was interpreted at the 5% significance level
Statistical Analysis 2: Comparison: Risperidone LAI; Within-group comparison of the change from baseline to endpoint in total PANSS score. The endpoint of the study was based on the LOCF principle; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 3: Comparison: Quetiapine; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.1026, Wilcoxon signed-rank test — The statistical test was interpreted at the 5% significance level

4. Secondary Outcome: Change From Baseline to Endpoint in Clinical Global Impression Scale (CGI) Score
Description: The 7-point CGI scale of Severity (CGI-S) was used to assess the severity of a subject's psychotic condition (0= normal, not at all ill, 1= borderline, etc. and 6= among the most extremely ill subjects).
Time Frame: Assessed at each visit from the moment the subject was randomized to a treatment arm (baseline visit) until the end of treatment (Month 24 or earlier)
Population: Efficacy analysis set, defined as all subjects who received at least 1 dose of study medication and had at least 1 efficacy assessment after baseline. This excluded 2 subjects of the risperidone LAI arm, 11 of the quetipaine arm, and 1 of the aripiprazole arm. One additional subject in the risperidone LAI arm did not have CGI data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone LAI | Quetiapine | Aripiprazole
Number analyzed (Participants) | 326 | 326 | 44
units on a scale | -0.3 (1.25) | 0.1 (1.24) | -0.1 (1.32)
Statistical Analysis 1: Comparison: Risperidone LAI vs Quetiapine; Between-group comparison of the change from baseline to endpoint in CGI-S score. The endpoint of the study was based on the LOCF principle; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — The statistical test was interpreted at the 5% significance level
Statistical Analysis 2: Comparison: Risperidone LAI; Within-group comparison of the change from baseline to endpoint in CGI-S score. The endpoint of the study was based on the LOCF principle; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 3: Comparison: Quetiapine; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.0446, Wilcoxon signed-rank test — The statistical test was interpreted at the 5% significance level

5. Secondary Outcome: Change From Baseline to Endpoint in Short-Form Health Survey 12 (SF-12) Scores
Description: Quality of life was assessed by means of the 12-item SF-12® survey. Two parameters, i.e., PCS (physical component summary) and MCS (mental component summary) were calculated. Both components scores range from 0 to 100 with higher scores indicating better QOL.
Time Frame: Assessed at the moment the subject was randomized to a treatment arm (baseline visit) and after 1, 3, 6, 12, 18, and 24 months of treatment
Population: Efficacy analysis set, defined as all subjects who received at least 1 dose of study medication and had at least 1 efficacy assessment after baseline. This excluded 2 subjects of the risperidone LAI, 11 of the quetipaine, and 1 of the aripiprazole arm. An additional 32, 32, and 2 subjects in the respective arms did not have SF-12 data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone LAI | Quetiapine | Aripiprazole
Number analyzed (Participants) | 295 | 294 | 42
units on a scale
  PCS score | 2.1 (9.04) | 1.0 (9.31) | 2.4 (10.36)
  MCS score | 3.2 (10.43) | 2.7 (10.88) | 4.9 (12.10)
Statistical Analysis 1: Comparison: Risperidone LAI vs Quetiapine; Between-group comparison of the change from baseline to endpoint in PCS score. The endpoint of the study was based on the LOCF principle; Test type: Superiority or Other; p = 0.0941, Wilcoxon (Mann-Whitney) — The statistical test was interpreted at the 5% significance level
Statistical Analysis 2: Comparison: Risperidone LAI; Within-group comparison of the change from baseline to endpoint in PCS score. The endpoint of the study was based on the LOCF principle; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 3: Comparison: Quetiapine; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.1146, Wilcoxon signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 4: Comparison: Risperidone LAI vs Quetiapine; Between-group comparison of the change from baseline to endpoint in MCS score. The endpoint of the study was based on the LOCF principle; Test type: Superiority or Other; p = 0.5589, Wilcoxon (Mann-Whitney) — The statistical test was interpreted at the 5% significance level
Statistical Analysis 5: Comparison: Risperidone LAI; Within-group comparison of the change from baseline to endpoint in MCS score. The endpoint of the study was based on the LOCF principle; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 6: Comparison: Quetiapine; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed-rank test — The statistical test was interpreted at the 5% significance level

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring between the first study-related procedure, i.e. screening visit, and 6 weeks after the last injection of risperidone LAI or the last intake of quetiapine or aripiprazole (24 months after baseline) were reported.
Description: AEs described hereafter are treatment-emergent AEs, defined as AEs that were new in onset or aggravated in severity following treatment start.
Arm/Group | Risperidone LAI | Quetiapine | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 63/329 | 77/337 | 7/45
Other Adverse Events (participants affected / at risk) | 201/329 | 213/337 | 28/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone LAI (N=329) | Quetiapine (N=337) | Aripiprazole (N=45)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abnormal behavior (Psychiatric disorders) | 0 | 1 | 0
Acquired methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 2 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 3 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Anal fistula (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 5 | 0
Asthenia (General disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 2 | 1 | 0
Condition aggravated (General disorders) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cyst removal (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1
Delusion (Psychiatric disorders) | 1 | 4 | 1
Depression (Psychiatric disorders) | 2 | 3 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Disturbance in social behavior (Psychiatric disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Drug level decreased (Investigations) | 0 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Family stress (Social circumstances) | 1 | 0 | 0
Gastic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lung injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 2 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Panic disorder (Psychiatric disorders) | 2 | 0 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 8 | 14 | 2
Refractory anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 2 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 7 | 0
Schizophrenia (Psychiatric disorders) | 14 | 23 | 0
Schizophrenia, disorganized type (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 4 | 4 | 0
Self injurious behavior (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Social problem (Social circumstances) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 5 | 1 | 0
Suicide attempt (Psychiatric disorders) | 5 | 2 | 0
Surgery (Surgical and medical procedures) | 1 | 0 | 0
Suspiciousness (Psychiatric disorders) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone LAI (N=329) | Quetiapine (N=337) | Aripiprazole (N=45)
Anxiety (Psychiatric disorders) | 39 | 30 | 7
Asthenia (General disorders) | 2 | 11 | 3
Delusion (Psychiatric disorders) | 4 | 4 | 4
Depression (Psychiatric disorders) | 15 | 16 | 3
Dizziness (Nervous system disorders) | 2 | 15 | 4
Headache (Nervous system disorders) | 19 | 16 | 5
Hyperprolactinaemia (Endocrine disorders) | 43 | 5 | 0
Insomnia (Psychiatric disorders) | 36 | 31 | 11
Nausea (Gastrointestinal disorders) | 1 | 6 | 5
Schizophrenia (Psychiatric disorders) | 4 | 17 | 0
Sleep disorder (Psychiatric disorders) | 8 | 2 | 3
Somnolence (Nervous system disorders) | 6 | 38 | 0
Tension (Psychiatric disorders) | 14 | 14 | 3
Weight decreased (Investigations) | 1 | 6 | 3
Weight increased (Investigations) | 23 | 20 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days